CLINICAL TRIAL: NCT05445284
Title: Group Education Trial to Improve Transition for Parents of Adolescents With Type 1 Diabetes: A Pilot Randomized Controlled, Superiority Trial (GET-IT For Parents)
Brief Title: Group Education Trial to Improve Transition for Parents of Adolescents With T1D
Acronym: GETIT-Parent
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Meranda Nakhla, Associate Professor, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-8592
Record Dates: First submitted 2022-06-27; First posted 2022-07-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Transition care; Pediatric; Adolescent; Parent; Education; Self-management; Hemaglobin A1c; Feasibility; Pilot randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Active arm: Participants randomized to the active arm will be asked to attend ≥ 3 group education sessions for parents of adolescents with T1D, in addition to their usual diabetes clinic visits every 3 months, over the 12-month intervention period. Group education sessions will coincide with regularly scheduled clinic visits.
  Control arm: Participants randomized to usual care will attend their usual 3-month interval diabetes clinic visits, over the 12-month intervention period, which consists of visits with their diabetes care physician.
Who Masked: Outcomes Assessor
Masking Description: Data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group education sessions for parents plus usual diabetes care (Experimental): ≥3 in-person/virtual one-hour group education sessions for parents plus usual diabetes care, every 3 months for 12 months and ≥3 "check-in" virtual 15-20 minute sessions in-between the group sessions. Each group session (3-8 parents per group) will be facilitated by a diabetes social worker and will consist of parent-driven discussions on topics relevant to adolescence and transition care. Each one-hour session will commence with an ice-breaker activity and then move to a parent-driven, facilitator-mediated discussion. The group session content will be guided by the needs of the participants; however, the facilitator will actively promote discussion on adolescent- and transition-related topics. The group discussion will end with participants setting goals for their next session.
  Interventions: Behavioral: Group education sessions for parents plus usual diabetes care
- Usual diabetes care (Other): Usual diabetes care, every 3 months for 12 months, which consists of visits with their diabetes care physician. In addition, as per usual care, individual sessions and meetings related to transition care with the diabetes social worker will be provided to parents, as needed.
  Interventions: Other: Usual diabetes care

INTERVENTIONS:
Behavioral: Group education sessions for parents plus usual diabetes care — ≥3 in person/virtual group education sessions for parents in addition to usual diabetes care, every 3 months for 12 months
  Arms: Group education sessions for parents plus usual diabetes care
Other: Usual diabetes care — Usual diabetes care, every 3-month for 12 months
  Arms: Usual diabetes care

SUMMARY:
The investigators will study if group education for parents of adolescents with type 1 diabetes (T1D) will improve the transition from adolescence to adulthood. The investigators aim to conduct a pilot randomized controlled trial (RCT) of parent group education sessions to assess the feasibility and refine the intervention to inform a full-scale multicenter RCT. The aims of the pilot are to estimate: 1. Recruitment rate, 2. Adherence rate, 3. Response rate, and 4. Retention rate. The aims for the future full-scale multicenter RCT are to assess the effect of parent group education sessions integrated into pediatric care, compared with usual care on self-management, hemoglobin A1c (HbA1c), adverse outcomes and validated measures during the transition from adolescence to adulthood. The investigators will conduct a parallel group, blinded (outcome assessors, data analysts), superiority pilot RCT of parents and their adolescents with T1D (14-16 years of age) followed at a university teaching hospital-based pediatric diabetes clinic in Montreal. Interventions will occur over 12-months. Follow-up will be to 18 months from enrollment.

DETAILED DESCRIPTION:
Rationale. Adolescence is a challenging life stage that is complicated for those with type 1 diabetes (T1D) as they learn to take responsibility for their health. Parents face uncertainty of what constitutes appropriate involvement and express distress around the health consequences of transferring responsibility to their adolescent. We know little about how to provide transition care services to parents as they attempt to support their adolescents during the transition to adulthood. We are currently conducting a multicenter randomized controlled trial (RCT) evaluating patient-driven group education for adolescents with T1D. Parents have expressed a need for education on how to transition responsibility of diabetes care from parent to adolescent. The investigators propose to study if group education for parents of adolescents with T1D will improve the transition from adolescence to adulthood. The investigators will conduct a pilot RCT of parent group education sessions to assess the feasibility and refine the intervention for a full-scale multicenter RCT.

Aims. The aims of the pilot are to estimate: 1. Recruitment rate, 2. Adherence rate, 3. Response rate, and 4. Retention rate. Through semi-structured interviews with parents, we also aim to identify aspects of the intervention that require refinement for the future full-scale multicenter RCT (e.g. session content and format). To assess feasibility success, we propose the following criteria:1. Recruitment rate: At least 50% of approached parents/adolescents will agree to randomization; 2. Adherence rate: At least 80% of parents attend ≥3 group education sessions; 3. Response rate: At least 80% of parents and adolescents will complete all validated questionnaires; 4. Retention rate: At least 70% of parents and adolescents will complete the trial. The aims for the future full-scale multicenter RCT are to determine the impact of parent group education sessions, compared with usual care on self-management, HbA1c, number of T1D-related emergency department visits and hospitalizations, diabetes distress, family conflict, diabetes resilience and diabetes responsibility.

Methods. The investigators will conduct a parallel group, blinded (outcome assessors, data analysts), superiority pilot RCT of parents and their adolescents with T1D (14-16 years of age) followed at a university teaching hospital-based pediatric diabetes clinic in Montreal. Dyads of adolescents and one parent will be recruited over 12 months. Interventions will occur over 12-months. Follow-up will be to 18 months from enrollment. Allocation will be concealed with a 1:1 intervention to control ratio. Visits in the active arm will consist of a parent group education session plus usual diabetes care every 3 months. The parent group education session, facilitated by a diabetes social worker, will consist of a parent-driven, in-person/virtual discussion on topics relevant to adolescence and transition care. Control arm participants will have usual care with their diabetes care provider every 3 months. Pilot RCT results will inform modification of trial execution related to feasibility and intervention for full-scale multicenter RCT. Main outcome measures are descriptions of study feasibility parameters. Health-related outcomes as well as parent and adolescent reported outcomes, using validated self-administered questionnaires will also be collected at baseline, 6, 12 and 18 months. Parents will be interviewed at baseline and 18 months to explore parents' experiences with and perceptions of the accessibility, acceptance, and usefulness of parent group education content and format, using qualitative descriptive methodology. Analysis will be descriptive and baseline data will be summarized, separately for those in the active and control arms.

ELIGIBILITY:
Inclusion Criteria:

* Parents and their adolescents, ages 14-16 years, with a diagnosis of T1D, of at least 6-months. Parent is defined as mother, father, or primary caregiver.
* Receiving diabetes care at a university teaching hospital-based pediatric diabetes clinic in Montreal: Montreal Children's Hospital (MCH)
* Participants must be fluent in English or French

Exclusion Criteria:

* Severe neurocognitive disabilities that may preclude parent's ability to participate in a group session
* Parents of adolescents participating in the Group Education Trial to Improve Transition in Type 1 Diabetes (GET-IT-T1D) for adolescents

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 12 months
  Recruitment rate. Proportion of all parents/adolescents approached agreeing to randomization. Feasibility success criteria: at least 50% of approached parents/adolescents agree to participate
Adherence feasibility | 12 months
  Adherence rate. Proportion of randomized parents attending ≥3 group education sessions. Feasibility success criteria: at least 80% of parents attend at least 3 one-hour group education/support sessions
Response feasibility | 18 months
  Response rate. Proportion of parents and adolescents completing all validated questionnaires. Feasibility success criteria: at least 80% parents/adolescents complete all questionnaires
Retention feasibility | 18 months
  Retention rate. Proportion of parents/adolescents completing the 18-month outcome measures. Feasibility success criteria: at least 70% of parents/adolescents complete the trial

SECONDARY OUTCOMES:
Parent group education session accessibility, acceptance, usefulness | 0, 18 months
  Parent interviews to explore parents' experiences with and perceptions of the accessibility, acceptance, and usefulness of the parent group education content and format, using qualitative descriptive methodology
Self-Management | 0, 6, 12, 18 months
  Self-Care Inventory-Revised Questionnaire assesses parent and adolescent self-management. The scores range from 1 to 5. Items scores are averaged to compute the score. A higher score represents a better outcome.
Diabetes Distress - Adolescent | 0, 6, 12, 18 months
  Problem Areas in Diabetes Scale-Teen (PAID-T) assesses adolescent diabetes distress. The scores range from 14 to 84. A total distress score is computed by summing responses. Higher scores indicate youth perception of feeling more burdened related to T1D.
Diabetes Distress - Parent | 0, 6, 12, 18 months
  Problem Areas in Diabetes Scale-Parent (PAID-P) assesses parent diabetes distress. The scores range from 15 to 90. A total distress score is computed by summing responses. Higher scores indicate higher levels of distress and burden.
Family Conflict | 0, 6, 12, 18 months
  Diabetes Family Conflict Scale assesses parent and adolescent family conflict. Total scores range from 19 to 57. A total score is calculated by summing all the item scores. Higher scores reflect greater family conflict.
Diabetes Resilience - Adolescent | 0, 6, 12, 18 months
  DSTAR-youth assesses adolescent diabetes resilience. Total scores range from 12 to 60. A total score is calculated by summing all the item scores. Higher scores reflect greater diabetes resilience.
Diabetes Resilience - Parent | 0, 6, 12, 18 months
  Diabetes-Specific Self-Compassion Scale assesses parent diabetes resilience. The score ranges from 1 to 5. A total score is calculated by reverse-scoring the 11 negatively-worded items and taking the mean of all items. Higher scores indicate greater diabetes-specific self compassion.
Responsibility (DFRQ) | 0, 6, 12, 18 months
  Diabetes Family Responsibility Questionnaire (DFRQ) assesses parent and adolescent responsibility (tasks in the family that contribute to the adolescent's diabetes management). Responsibilities are reflected in three domains: general health maintenance, regimen tasks, and social presentation. A total mean score across items is calculated. The score ranges from 1 to 3. Higher scores reflect that the adolescent is taking or initiating responsibility almost all the time.
Responsibility (RCBRS) | 0, 6, 12, 18 months
  Readiness to Change the Balance of Responsibility Scale (RCBRS) assesses parent and adolescent responsibility. The score ranges from 1 to 5. A mean score of the 12 items (parent) and the seven items (youth) is calculated. Higher scores represent more readiness to change.
Hemaglobin A1c (HbA1c) | 0, 6, 12, 18 months
  HbA1c is measured at each pediatric diabetes care visit every 3 months as part of the standard of diabetes care and is measured with a capillary blood sample using point of care testing (DCA 2000).HbA1c will be identified from medical record chart.
Diabetes-related hospitalizations | 0, 12 months
  Any diabetes-related hospitalizations in the past 12 months, expressed as number of hospitalizations per person-years (P-Y) at risk will be derived from medical record chart.
Diabetes-related emergency department visits | 0, 12 months
  Any diabetes-related emergency-department visits in the past 12 months, expressed as number of emergency department visits per person-years (P-Y) at risk will be derived from medical record chart

CONTACTS AND LOCATIONS:
Overall Officials: Meranda Nakhla, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital - McGill University Health Centre (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data supporting the results reported in the published research articles, after de-identification will be available only for the full-scale RCT.

REFERENCES:
- [Background] Ladd JM, Reeves-Latour J, Dasgupta K, Bell LE, Anjachak N, Nakhla M. Toward a better understanding of transition from paediatric to adult care in type 1 diabetes: A qualitative study of adolescents. Diabet Med. 2022 May;39(5):e14781. doi: 10.1111/dme.14781. Epub 2022 Jan 7. PMID 34967058
- [Background] Alwadiy F, Mok E, Dasgupta K, Rahme E, Frei J, Nakhla M. Association of Self-Efficacy, Transition Readiness and Diabetes Distress With Glycemic Control in Adolescents With Type 1 Diabetes Preparing to Transition to Adult Care. Can J Diabetes. 2021 Jul;45(5):490-495. doi: 10.1016/j.jcjd.2021.05.006. Epub 2021 May 19. PMID 34176613
- [Background] Robinson ME, Simard M, Larocque I, Shah J, Rahme E, Nakhla M. Psychiatric disorders in emerging adults with diabetes transitioning to adult care: A retrospective cohort study. Diabet Med. 2021 Jun;38(6):e14541. doi: 10.1111/dme.14541. Epub 2021 Feb 19. PMID 33576092
- [Background] Mok E, Henderson M, Dasgupta K, Rahme E, Hajizadeh M, Bell L, Prevost M, Frei J, Nakhla M. Group education for adolescents with type 1 diabetes during transition from paediatric to adult care: study protocol for a multisite, randomised controlled, superiority trial (GET-IT-T1D). BMJ Open. 2019 Nov 11;9(11):e033806. doi: 10.1136/bmjopen-2019-033806. PMID 31719096
- [Background] Michaud S, Dasgupta K, Bell L, Yale JF, Anjachak N, Wafa S, Nakhla M. Adult care providers' perspectives on the transition to adult care for emerging adults with Type 1 diabetes: a cross-sectional survey. Diabet Med. 2018 Jul;35(7):846-854. doi: 10.1111/dme.13627. Epub 2018 May 2. PMID 29577410
- [Background] Nakhla M, Bell LE, Wafa S, Dasgupta K. Improving the transition from pediatric to adult diabetes care: the pediatric care provider's perspective in Quebec, Canada. BMJ Open Diabetes Res Care. 2017 Jun 30;5(1):e000390. doi: 10.1136/bmjdrc-2017-000390. eCollection 2017. PMID 28761657
- [Background] Wafa S, Nakhla M. Improving the Transition from Pediatric to Adult Diabetes Healthcare: A Literature Review. Can J Diabetes. 2015 Dec;39(6):520-8. doi: 10.1016/j.jcjd.2015.08.003. Epub 2015 Oct 20. PMID 26498219
- [Background] Nakhla M, Daneman D, To T, Paradis G, Guttmann A. Transition to adult care for youths with diabetes mellitus: findings from a Universal Health Care System. Pediatrics. 2009 Dec;124(6):e1134-41. doi: 10.1542/peds.2009-0041. Epub 2009 Nov 23. PMID 19933731
- [Background] Nakhla M, Daneman D, Frank M, Guttmann A. Translating transition: a critical review of the diabetes literature. J Pediatr Endocrinol Metab. 2008 Jun;21(6):507-16. PMID 18717235
- [Derived] Tapp K, Mok E, Davis D, Guerin-Marion S, Frei J, Gibbon M, Henderson M, Miljanovski M, Da Costa D, Shulman R, Nakhla M, Kichler J. Perspectives of parents/caregivers prior to a pilot intervention trial to improve transition to adult care for adolescents with type 1 diabetes: A qualitative study. BMJ Open. 2025 Dec 29;15(12):e108079. doi: 10.1136/bmjopen-2025-108079. PMID 41469044